CLINICAL TRIAL: NCT05875506
Title: Efficacy of Ozone Gel, Doxycycline Saturated Chitosan Dressing Versus Alveogyl in Pain Alleviation and Healing of Alveolar Osteitis in Diabetic Patients Double Blind Randomized Clinical Trial
Brief Title: Efficacy of Ozone Gel, Doxycycline Saturated Chitosan Dressing Versus Alveogyl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Tarek Abdelbarry, Lecturer of Oral and Maxillofacial Surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 713
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2023-05

CONDITIONS: Osteitis; Dry Socket
MeSH Terms: conditions — Osteitis; Dry Socket

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ozone gel (Experimental): (Ozene; Premier Research Labs, lp, 3500-b Wadley pl, Austin, TX, USA. 78728)
  Interventions: Drug: Ozone gel
- doxycycline hyclate saturated chitosan dressing (Experimental): doxycycline hyclate ( Atridox 10% Tolmar Inc, USA) saturated chitosan dressing (HHD) HemCon dental dressing Pro ( Tricol Biomedical, Inc. USA)
  Interventions: Drug: doxycycline hyclate saturated chitosan dressing
- Alveogyl paste (Active Comparator): Alveogyl paste ( Septodont, inc, france)
  Interventions: Drug: Ozone gel; Drug: doxycycline hyclate saturated chitosan dressing

INTERVENTIONS:
Drug: Ozone gel — (Ozene; Premier Research Labs, lp, 3500-b Wadley pl, Austin, TX, USA. 78728) applied in dry socket
  Arms: Alveogyl paste; Ozone gel
Drug: doxycycline hyclate saturated chitosan dressing — doxycycline hyclate ( Atridox 10% Tolmar Inc, USA) saturated chitosan dressing (HHD) HemCon dental dressing Pro ( Tricol Biomedical, Inc. USA) applied in dry socket
  Arms: Alveogyl paste; doxycycline hyclate saturated chitosan dressing

SUMMARY:
Efficacy of ozone gel, doxycycline saturated chitosan dressing versus Alveogyl in pain alleviation and healing of alveolar osteitis in diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20 years and under 60 years of age
* DM controlled by medication, presented to outpatient clinic with signs and symptoms of dry socket
* Only participant that are willing to control and record blood glucose level throughout the study period

Exclusion Criteria:

* Patients with any significant medical condition (besides DM)
* Alcoholic individuals
* Patients on drugs that affect the central nervous systems
* Patients who reported the use of drugs that might interfere with pain sensitivity
* Pregnant and lactating women
* Hypersensitivity to local anesthetics

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Pain scores will be recorded on visual analog scale (VAS) | 7 days
  visual analog scale (VAS) is a scale from 0 to 10. 0 indicates no pain while indicates extensive unbearable pain

SECONDARY OUTCOMES:
Healing score of the extraction socket | 21 days
  According to the amount of granulation tissue:
  Nil: no granulation tissue
  * Granulation tissue in one quarter or less
    * Granulation tissue in 2 quarters +++ Granulation tissue in 3 quarters ++++ Granulation tissue in 4 quarters

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No